CLINICAL TRIAL: NCT06895824
Title: Can Somatic Tracking Help People Living with Tinnitus?
Brief Title: Somatic Tracking for Tinnitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University College London Hospitals (Other)
Responsible Party: Principal Investigator, Dr Florian Vogt, Consultant Clinical Psychologist, Head of Department of Clinical Psychology, Audiovestibular Medicine, University College London Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21415/001
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Tinnitus
Keywords: tinnitus; mindfulness; mindfulness meditation; somatic tracking; tinnitus distress
MeSH Terms: conditions — Tinnitus | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Intervention group participants will be given the choice to proceed to the Tinnitus Tracking [TT] intervention, a 15-minute somatic tracking guided meditation recorded by Dr Florian Vogt, a tinnitus treatment specialist, immediately or the next day. Before starting the first session of the TT intervention, participants answer the question, 'Right now, how annoying is your tinnitus?" using ratings on a scale from 1 (not at all) to 10 (much more). Each session of the TT intervention involves the guided meditation session, followed by the tinnitus annoyance rating. Participants will be reminded to complete one session daily over a period of two weeks and will only be allowed to access the experiment once a day. Reminders will be sent daily via email by Gorilla, once access to the intervention for the day has been provided.
  Interventions: Other: Mindfulness Meditation
- Control (No Intervention): Participants in this arm do not have tasks to complete over the two-week study period. A wait-list control condition will be set-up for this group, whereby participants will receive the intervention after completing the follow-up measures in two weeks. Since our sample is non-clinical and less at risk, we believe the two week delay period should not cause distress or adverse events.

INTERVENTIONS:
Other: Mindfulness Meditation — Somatic tracking is one aspect of most mindfulness meditation protocols, involving paying attention to the present non-judgementally, and focusing on breath and bodily sensations (e.g., sounds in the case tinnitus). This study employs this approach as a standalone intervention, in the form of a guided meditation recording.
  Other Names: Somatic Tracking
  Arms: Intervention

SUMMARY:
We are examining the effect of mindfulness meditation on attitudes towards tinnitus, as well as physical and psychological distress associated with the condition. The meditation is designed to promote neuroplasticity, fostering new neural connections to help you reinterpret tinnitus through a lens of safety and reduce the perception of threat. This approach integrates several techniques from various psychological therapies which have been promising in reducing tinnitusrelated distress. Therefore, the purpose of this study is to see whether a guided mindfulness meditation intervention is effective in improving the acceptance of tinnitus symptoms, as well as reducing tinnitus-related distress in people living with tinnitus.

DETAILED DESCRIPTION:
Somatic tracking is one aspect of most mindfulness meditation protocols, involving paying attention to the present non-judgementally, and focusing on breath and bodily sensations (e.g., sounds in the case tinnitus). By encouraging individuals to observe and reinterpret distressing symptoms as benign, it aims to decrease the brain's reactivity and vigilance towards tinnitus symptoms, promoting acceptance instead of maladaptive avoidance behaviours that can inadvertently heighten awareness of symptoms (McKenna et al., 2020). Reduced tinnitus-related fear has appeared to improve CBT treatment effects (Cima et al., 2018), while greater tinnitus acceptance is associated with reduced tinnitus distress and improved mental well-being (Westin et al., 2008). This coping strategy has also reduced distress in other conditions, such as traumatic brain injury (Garland et al., 2009). In line with the greater goals of mindfulness, somatic tracking encourages sustained and flexible attention to the wider experience and environment, moving away from narrowed attention to tinnitus symptoms. In redeploying attention beyond tinnitus, awareness extends to other stimuli, and tinnitus-related distress should reduce alongside decreased resistance and selective attention which contribute to the perception of tinnitus (Marks et al., 2020b). This study aims to explore the effectiveness of a somatic tracking intervention - Tinnitus Tracking, for tinnitus sufferers. This intervention constitutes a mindfulness activity commonly part of meditation/mindfulness programmes, which will be tested as a standalone intervention. We aim to answer: What is the effect of Tinnitus Tracking compared to no intervention on (1) participants' positive and negative thoughts towards their tinnitus and (2) the physical and psychological distress associated with the condition?

ELIGIBILITY:
Inclusion Criteria:

* Experiencing distressing tinnitus
* Sufficient English language and hearing ability to take part
* Completed all relevant medical and audiological investigations and concluded ensuing treatment for any underlying disease
* Not be engaging in any other therapy for tinnitus.

Exclusion Criteria:

* Risk to self (scoring 'nearly every day' on PHQ-9 question "Thoughts that you would be better off dead, or of hurting yourself in some way?")
* Severe mental health difficulties (PHQ-9 score of 20 or more)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-11 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Cognitions about Tinnitus | Baseline and 2 weeks
  Positive and negative thoughts about tinnitus will be assessed with the Tinnitus Cognitions Questionnaire (TCQ) (Wilson & Henry 1998). It consists of 26 items (statements) rated on a 5-point Likert scale. For example, "if only the noise would go away." The first 13 items refer to negative thoughts and the second 13 items refer to positive thoughts. The TCQ has been supported as a valid measure of positive and negative thinking in tinnitus (Handscomb et al., 2017), demonstrates good reliability, and is suitable for research use
Psychological Distress | Baseline and 2 weeks
  Depression will be assessed on the Patient Health Questionnaire-9 (PHQ-9) (Kroenke et al., 1999), with nine items, such as "Feeling down, depressed, or hopeless?". Anxiety will be assessed on the Generalised Anxiety Disorder Assessment-7 (GAD-7) (Spitzer et al., 2006), with seven items, for example "Feeling afraid as if something awful might happen". Both the PHQ-9 and GAD-7 have been shown to be valid and reliable in assessing depressive and anxious symptoms respectively.
Tinnitus Severity | Baseline and 2 weeks
  Tinnitus severity will be assessed using the Tinnitus Functional Index (TFI) (Meikle et al., 2012). It consists of 25 items covering overall tinnitus severity and negative impact. The TFI has demonstrated sensitivity to treatment-related change, high validity, and good reliability. The measure has been concluded to be suitable for both clinical and research purposes.
Tinnitus Annoyance Rating | Baseline and daily over 2 weeks
  Participants answer the question, 'Right now, how annoying is your tinnitus?" using ratings on a scale from 1 (not at all) to 10 (much more). Each session of the TT intervention involves the guided meditation session, followed by the tinnitus annoyance rating.

SECONDARY OUTCOMES:
Post-Study Feedback | At the end of the study (2 weeks)
  Data from the post-study feedback survey, regarding satisfaction with and acceptability of the intervention and study.

CONTACTS AND LOCATIONS:
Locations (1):
- Online, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
After the research, all research documents (e.g. questionnaires, responses) will be securely stored on UCL's Research Data Storage System (RDSS). After data analysis and sharing of results with interested participants all identifiable data (i.e., email address) will be deleted.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Research documents/data will be kept on UCL's RDSS for one year. At the end of the one-year period, the data will be automatically deleted.